CLINICAL TRIAL: NCT06254794
Title: Effect of Blood Flow Restriction (BFR) Rehabilitation After Achilles Tendon Rupture Reconstruction
Brief Title: Effect of BFR Rehab After Achilles Tendon Rupture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, The John S. Dunn Chair in Orthopedic Surgery, Professor of Clinical Orthopedic Surgery, Vice-Chairman Dept. of Orthopedic Surgery, Head Team Physician: Rice University, Team Physician / Consultant: MLB, Houston Ballet, NASA Astronaut Corps., The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019305
Record Dates: First submitted 2023-12-22; First posted 2024-02-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Achilles Tendon Rupture
Keywords: achilles tendon rupture; blood flow restriction
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: The Delfi PTS device for BFR allows for a systematic and customized approach to BFR training in the clinic. This instrument provides a digital display of pressure, inflation time, and provides the user with an interface to control the tourniquet system. Pressure is monitored and regulated continuously to compensate for changing levels in the cuff during movement. Each cuff is specifically designed for the tapered contour of a body limb (arm or leg) and sized appropriately based on body region. These cuffs only work with the Delfi PTS device and allow for comfortable pressure application. Exercise will be performed with the cuff placed around the proximal limb and inflated through the duration of activity (~5 minutes), then immediately deflated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Blood flow restriction group (Experimental): The study group will undergo normal Achilles tendon rupture reconstruction rehab modified by use of a tourniquet for blood flow restriction during selected exercises.
  Interventions: Device: Blood flow restriction with Delfi Personalized Tourniquet System (PTS); Other: Physical therapy
- Standard of Care (control) group (Other): The control group will undergo the normal Achilles tendon rupture reconstruction rehab protocol as determined by Drs. Varner and McCulloch.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Device: Blood flow restriction with Delfi Personalized Tourniquet System (PTS) — Standard of care physical therapy exercises with the use of the Delfi PTS cuff
  Arms: Blood flow restriction group
Other: Physical therapy — Standard of care physical therapy exercises

SUMMARY:
The purpose of this study is to determine if blood flow restriction therapy after Achilles tendon rupture reconstruction decreases post-operative calf atrophy, improves reported outcomes, and ultimately decreases return to play time.

DETAILED DESCRIPTION:
The purpose of this research study is to determine if the use of Blood Flow Restriction, BFR, therapy in addition to standard physical therapy (PT) for post-Achilles tendon rupture reconstruction will decrease post-operative muscle atrophy (loss of muscle), increases dorsal and planar ankle flexion (range of motion), increase strength, and ultimately decrease return to play time for the BFR therapy group as compared to the control group.

Participants in this study will be randomly divided into either BFR group that will receive BFR therapy in addition to standard physical therapy protocol post-operatively or the control group which will undergo the standard PT protocol. All participants will complete full body composition scans (DEXA) and questionnaires before surgery, prior to physical therapy (three weeks post-op), eight weeks post-op, and 16 weeks post-op. Subjective and objective measures will be taken at physical therapy eight weeks and 16 weeks post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Achilles Rupture confirmed by MRI or Thompson Test
* Adult
* Receiving Percutaneous Achilles Repair System (PARS) or open repair
* Proposed PT with Methodist Location

Exclusion Criteria:

* Obesity (BMI>35)
* Diabetes
* Cardiovascular, renal, liver or pulmonary disease
* Active infections
* Cancer (current or treated within the past 2 years) or coagulation disorder
* Physically unable to participate in the intervention
* Unable to complete a minimum of 85% of the assigned rehabilitation sessions
* Less than 18 years of age
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2018-11-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Muscle mass preservation | pre-op, 4 weeks post op, 8 weeks post op, 16 weeks post-op
  Lean mass for lower extremity measured in kilograms (kg) using Dual-Energy-Xray-Absorptiometry (DEXA).
Bone density preservation | pre-op, 4 weeks post op, 8 weeks post op, 16 weeks post-op
  Bone mineral content measured in grams using Dual-Energy-Xray-Absorptiometry (DEXA).
Improve patient reported outcomes (Physical activity) | pre-op, 4 weeks post op, 8 weeks post op, 16 weeks post-op
  Digital RedCap survey tool sends Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function survey which consists of questions about their physical health and patient responds with Excellent, Very Good, Good, Fair or poor. Using healthmeasures.net, responses are converted to T-scores based on the general population. The highest the T-scores, the better physical health the patient has.
Improve patient reported outcomes (Pain) | pre-op, 4 weeks post op, 8 weeks post op, 16 weeks post-op
  Digital RedCap survey tool sends Pain Visual Analog Scale asking patients to rate their pain from 0 (no pain) to 100 (worst pain possible).
Improve patient reported outcomes (Achilles tendon survey) | pre-op, 4 weeks post op, 8 weeks post op, 16 weeks post-op
  Digital RedCap survey tool sends Achilles Tendon Rupture Score (ATRS) survey. This survey asks 10 questions where the patient answers from 0=major limitation to 10=No limitations. High scores point to better physical activity.
Change in range of motion | Starting 4 weeks post op, patient will go to physical therapy twice a week until week 16.
  Physical therapy will do functional assessments including: leg squat depth, Y balance anterior, y balance posteromedial, y balance posterolateral and measure in centimeters (cm). The measurements will be taken at each physical therapy appointment and compared at the end of the study.
Change in single heel raise repetitions | Starting 4 weeks post op, patient will go to physical therapy twice a week until week 16.
  Physical therapy will count how many heel raises can be done at each timepoint.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No